CLINICAL TRIAL: NCT04714359
Title: A Multi-Site Open-Label Safety Extension Study of Manualized MDMA-Assisted Psychotherapy for the Treatment of Participants With Posttraumatic Stress Disorder
Brief Title: A Multi-Site Open-Label Extension Study of MDMA-Assisted Psychotherapy for PTSD
Acronym: MAPPUSX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lykos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAPPUSX
Record Dates: First submitted 2021-01-14; First posted 2021-01-19 (Actual); Results first posted 2024-11-29 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MDMA-assisted therapy (Experimental): Three open-label sessions of MDMA-assisted therapy, each scheduled approximately 1 month apart, with initial dose of midomafetamine HCl of 80 or 120 mg and optional supplemental dose half that of initial dose (40 or 60 mg) 1.5 to 2 hours later
  Interventions: Drug: Midomafetamine HCl

INTERVENTIONS:
Drug: Midomafetamine HCl — Initial doses per Experimental Session include 80 mg or 120 mg midomafetamine HCl, followed 1.5 to 2 hours later by a supplemental dose unless tolerability issues emerge. For an initial dose of 80 mg, a 40 mg supplemental dose will be used. For an initial dose of 120 mg, a 60 mg supplemental dose will be used. Total amounts of midomafetamine HCl to be administered per Experimental Session range from 80 mg to 180 mg.
  Other Names: 3,4-methylenedioxymethamphetamine; MDMA HCl; midomafetamine; MDMA

SUMMARY:
The goal of this clinical trial is to learn if MDMA-assisted therapy is safe and effective at reducing PTSD symptoms in people with PTSD who received placebo in a prior MDMA-assisted therapy study.

The main question it aims to answer is:

Do PTSD symptoms decrease in people who receive a flexible dose of MDMA (120 or 180 mg MDMA HCl) with therapy in three sessions?

Participants will undergo three preparatory therapy sessions without any study drug, then three MDMA-assisted therapy sessions with a flexible dose of 80 or 120 mg, followed by three integrative therapy sessions without study drug after each MDMA-assisted therapy session.

DETAILED DESCRIPTION:
This multi-site, open-label safety extension study assesses the efficacy and safety of MDMA-assisted psychotherapy versus psychotherapy in participants diagnosed with PTSD. The study will be conducted in N ≈ 100 participants. Participants who were randomized to the placebo arm in either of the two parent Phase 3 trials of MDMA-assisted psychotherapy and who meet all other entry criteria will be eligible and invited to participate in this study. In addition, participants in the parent Phase 3 trials who were unable to complete the study due to the COVID-19 pandemic or other unforeseen circumstances may participate in this study.

The treatment consists of an initial dose of midomafetamine HCl (80 or 120 mg), followed by a supplemental dose (40 or 60 mg) unless contraindicated, administered with manualized psychotherapy in three open-label Experimental Sessions each spaced approximately one month apart. During Experimental Session 1, participants will receive an initial dose of 80 mg of midomafetamine HCl, followed by a supplemental dose of 40 mg. During Experimental Sessions 2 and 3, participants will receive an initial dose of 80 or 120 mg of midomafetamine HCl, followed by a supplemental dose of 40 or 60 mg.

This Treatment Period is preceded by three Preparatory Sessions. During the Treatment Period, each Experimental Session is followed by three Integrative Sessions of non-drug psychotherapy. Experimental Sessions are followed by an overnight stay, with the exception of a subset of participants who will be invited to participate in a sub-study to assess the feasibility of Experimental Sessions without overnight stay. The primary study endpoint is the change from baseline in PCL-5 (PTSD Checklist for DSM-5) scores from Visit 3 to Visit 16.

ELIGIBILITY:
Inclusion Criteria:

* Were previously enrolled in a parent study and (meet one of the following):

  1. At time of unblinding, their treatment assignment was to the placebo arm; or,
  2. Did not begin Experimental Sessions due to the COVID-19 global pandemic or other unforeseen circumstances;
  3. Completed fewer than three Experimental Sessions prior to Study Termination due to the COVID-19 global pandemic or other unforeseen circumstances.
* Are considered in good standing with the study site at which they enrolled in a parent study; if, in the opinion of the investigator, therapy team, and Medical Monitor, the participant was compliant with protocol requirements, even if they were unable to complete all study visits.
* Are at least 18 years old
* Are fluent in speaking and reading the predominantly used or recognized language of the study site
* Are able to swallow pills
* Agree to have study visits recorded, including Experimental Sessions, Independent Rater assessments, and non-drug psychotherapy sessions
* Must provide a contact (relative, spouse, close friend or other caregiver) who is willing and able to be reached by the investigators in the event of a participant becoming suicidal or unreachable.
* Must agree to inform the investigators within 48 hours of any medical conditions and procedures
* If of childbearing potential, must have a negative pregnancy test at study entry and prior to each Experimental Session, and must agree to use adequate birth control through 10 days after the last Experimental Session.
* Must not participate in any other interventional clinical trials during the duration of the study
* Agree to the following lifestyle modifications: comply with requirements for fasting and refraining from certain medications prior to Experimental Sessions.
* Must be willing to remain overnight at the study site after each Experimental Session and be driven home after, and commit to medication dosing, therapy, and study procedures.

Exclusion Criteria:

* Are not able to give adequate informed consent Have uncontrolled hypertension
* Have a marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 milliseconds [ms] in males and >460 ms in females corrected by Fridericia formula)
* Have a history of additional risk factors for Torsade de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
* Have evidence or history of significant medical disorders, such as myocardial infarction, cerebrovascular accident, or aneurysm
* Have symptomatic liver disease
* Have recent history of hyponatremia or hyperthermia
* Weigh less than 48 kilograms (kg)
* Are pregnant or nursing, or are of childbearing potential and are not practicing an effective means of birth control
* Have an active illicit or prescription drug substance use disorder within 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (11):
  - New School Research, Los Angeles, California
  - San Francisco Insight and Integration Center, San Francisco, California
  - UCSF, San Francisco, California
  - Aguazul-Blue Water Inc., Boulder, Colorado
  - Wholeness Center, Fort Collins, Colorado
  - Ray Worthy Psychiatry, New Orleans, Louisiana
  - Trauma Research Foundation, Boston, Massachusetts
  - NYU, New York, New York
  - New York Private Practice, New York, New York
  - Zen Therapeutic Solutions, LLC, Mt. Pleasant, South Carolina
  - University of Wisconsin - Madison, Madison, Wisconsin
- Canada (2):
  - Numinus, Vancouver, British Columbia
  - Numinus, Montreal, Quebec
- Israel (2):
  - Beer Yaakov Mental Health Center, Beer Yaaqov
  - Tel Hashomer, Tel Aviv

IPD SHARING:
Plan to Share IPD: Yes
We will share outcome data appearing in any published reports upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data and study-related documents will be available when the database has been locked and data has been unblinded.
Access Criteria: Interested persons should correspond with the central contact for the multisite study.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who were randomized to the placebo arm in the two parent Phase 3 trials and who meet all other entry criteria will be eligible and invited to participate in this open-label safety extension study.
Groups:
- MDMA-assisted Therapy: Three open-label sessions of MDMA-assisted therapy with flexible dose of midomafetamine HCl (80 or 120 mg) and optional supplemental dose of (40 or 60 mg), 1.5 to 2 hours later
  Midomafetamine HCl: Three sessions of MDMA-assisted therapy with flexible dose of midomafetamine HCl from 80 to 120 mg and optional supplemental dose half that of initial dose 1.5 to 2 hours later
Period: Overall Study
Arm/Group | MDMA-assisted Therapy
Started | 87
Completed | 78
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | MDMA-assisted Therapy
Number analyzed (Participants) | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (9.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 73
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 8
  White | 54
  More than one race | 9
  Unknown or Not Reported | 0
Education [Mean (Standard Deviation); unit: years] | 17.1 (2.34)
Trauma History [Count of Participants; unit: Participants]
  Veteran | 14
  Served in combat area | 10
  Multiple traumatic events | 65

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Visit 16 in PCL-5 Total Score
Description: The Post Traumatic Stress Disorder Checklist for DSM-5 (PCL-5) is a 20-item self-report questionnaire in which respondents indicate the presence and severity of PTSD symptoms, derived from the symptoms of PTSD per DSM-5. Participants indicate how much distress they have experienced in the last 2 weeks due to symptoms such as "Repeated, disturbing memories, thoughts, or images of a stressful experience from the past," "Trouble remembering important parts of a stressful experience from the past," and "Feeling irritable or having angry outbursts" on a five-point Likert-type scale (0=Not at all to 4=Extremely). The total severity score can range from 0 to 80 and lower scores indicate less PTSD symptoms.
Time Frame: Baseline enrollment to approximately 18 weeks later (Visit 16 occurs 24 to 32 days after Experimental Session 3)
Population: The primary outcome analysis (change from baseline) is based on the n=81 participants with PCL-5 data available at the primary outcome visit (Visit 16).
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | MDMA-assisted Therapy
Number analyzed (Participants) | 81
score on a scale | -14.92 [-18.05 to -11.79]

2. Secondary Outcome: Change From Baseline to Visit 16 in Sheehan Disability Scale (SDS) Total Score
Description: The SDS is a self-report assessment of functional impairment. The reporting period for the SDS refers to the past month. The items indicate degree of impairment in the domains of work/school, social life, and home life, with response options based on an eleven-point scale (0=not at all to 10=extremely), with higher scores indicating greater functional impairment.
Time Frame: Baseline enrollment to approximately 18 weeks later (Visit 16 occurs 24 to 32 days after Experimental Session 3)
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | MDMA-assisted Therapy
Number analyzed (Participants) | 71
score on a scale | -4.10 [-5.95 to -2.25]

ADVERSE EVENTS:
Time Frame: From baseline to end of follow up (approximately 18 weeks)
Groups:
- Pre-Treatment MDMA-Assisted Therapy: Adverse events that occur during the Preparatory Period prior to the first dose in the first MDMA-assisted therapy session.
- On Day 0, 1, or 2 MDMA-Assisted Therapy: Adverse events that occur on the day of or within two days following each MDMA-assisted therapy session.
- Treatment-Emergent Adverse Events MDMA-Assisted Therapy: Adverse events that occur during the Treatment Period from the first Experimental Session to the last Integrative Session.
- Follow-Up MDMA-Assisted Therapy: Adverse Events that occurred after the last Integrative Session through follow-up.
Arm/Group | Pre-Treatment MDMA-Assisted Therapy | On Day 0, 1, or 2 MDMA-Assisted Therapy | Treatment-Emergent Adverse Events MDMA-Assisted Therapy | Follow-Up MDMA-Assisted Therapy
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/85 | 0/85 | 0/85
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/85 | 3/85 | 1/85
Other Adverse Events (participants affected / at risk) | 51/85 | 84/85 | 84/85 | 15/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-Treatment MDMA-Assisted Therapy (N=85) | On Day 0, 1, or 2 MDMA-Assisted Therapy (N=85) | Treatment-Emergent Adverse Events MDMA-Assisted Therapy (N=85) | Follow-Up MDMA-Assisted Therapy (N=85)
Abdominal sepsis (Infections and infestations) | NA | NA | 1 | 0
Colonic abscess (Infections and infestations) | NA | NA | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | NA | NA | 1 | 0
Diverticulitis (Infections and infestations) | NA | NA | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | NA | NA | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | NA | NA | 1 | 0
Retinal detachment (Eye disorders) | NA | NA | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-Treatment MDMA-Assisted Therapy (N=85) | On Day 0, 1, or 2 MDMA-Assisted Therapy (N=85) | Treatment-Emergent Adverse Events MDMA-Assisted Therapy (N=85) | Follow-Up MDMA-Assisted Therapy (N=85)
Palpitations (Cardiac disorders) | 0 | 7 | 7 | 0
Mydriasis (Eye disorders) | 0 | 13 | 13 | 0
Photophobia (Eye disorders) | 0 | 3 | 4 | 0
Nausea (Gastrointestinal disorders) | 4 | 33 | 38 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 16 | 16 | 0
Vomiting (Gastrointestinal disorders) | 0 | 10 | 13 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 4 | 7 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 7 | 7 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 4 | 5 | 0
Fatigue (General disorders) | 1 | 20 | 32 | 2
Therapeutic response unexpected (General disorders) | 2 | 23 | 24 | 0
Feeling hot (General disorders) | 0 | 19 | 19 | 0
Feeling cold (General disorders) | 1 | 16 | 16 | 0
Feeling abnormal (General disorders) | 2 | 9 | 12 | 0
Feeling of body temperature change (General disorders) | 0 | 12 | 12 | 0
Chills (General disorders) | 0 | 10 | 11 | 0
Feeling of relaxation (General disorders) | 1 | 8 | 8 | 0
Feeling jittery (General disorders) | 0 | 5 | 5 | 0
Gait disturbance (General disorders) | 0 | 5 | 5 | 0
Pain (General disorders) | 1 | 2 | 5 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 7 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 32 | 32 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 50 | 50 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 5 | 12 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 7 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 5 | 7 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 7 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 6 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 4 | 5 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 5 | 5 | 0
Headache (Nervous system disorders) | 7 | 43 | 49 | 1
Dizziness (Nervous system disorders) | 1 | 19 | 20 | 1
Nystagmus (Nervous system disorders) | 0 | 20 | 20 | 0
Paraesthesia (Nervous system disorders) | 0 | 17 | 18 | 0
Tremor (Nervous system disorders) | 0 | 9 | 10 | 0
Disturbance in attention (Nervous system disorders) | 1 | 5 | 6 | 1
Balance disorder (Nervous system disorders) | 0 | 5 | 5 | 0
Insomnia (Psychiatric disorders) | 4 | 25 | 33 | 0
Suicidal ideation (Psychiatric disorders) | 14 | 10 | 32 | 7
Anxiety (Psychiatric disorders) | 6 | 23 | 27 | 0
Depressed mood (Psychiatric disorders) | 2 | 14 | 20 | 0
Bruxism (Psychiatric disorders) | 0 | 11 | 11 | 0
Restlessness (Psychiatric disorders) | 1 | 9 | 11 | 0
Emotional disorder (Psychiatric disorders) | 0 | 7 | 10 | 2
Anger (Psychiatric disorders) | 1 | 6 | 8 | 0
Depression (Psychiatric disorders) | 0 | 3 | 8 | 0
Nightmare (Psychiatric disorders) | 4 | 5 | 7 | 0
Panic attack (Psychiatric disorders) | 2 | 5 | 7 | 0
Irritability (Psychiatric disorders) | 1 | 2 | 5 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 7 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 7 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 24 | 24 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (3):
  • Study Protocol (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/59/NCT04714359/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-13): https://cdn.clinicaltrials.gov/large-docs/59/NCT04714359/SAP_001.pdf
  • Informed Consent Form (2023-05-04): https://cdn.clinicaltrials.gov/large-docs/59/NCT04714359/ICF_002.pdf